CLINICAL TRIAL: NCT00322257
Title: Inhaled Mealtime Insulin With the AERx® iDMS Versus Subcutaneous Injected Insulin Aspart Both in Combination With Insulin Detemir in Type 1 Diabetes: A 104 Week, Open-Label, Multicenter, Randomised, Parallel Trial (Followed by a Twelve-Week Re-Randomised Extension) To Investigate Safety and Efficacy
Brief Title: Safety and Efficacy of Inhaled Insulin in Type 1 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-2076
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: inhaled human insulin; Drug: insulin detemir
- B (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Arms: A
Drug: insulin detemir — Injection s.c., 50% of daily dose
  Other Names: Levemir, NN304
Drug: insulin aspart — Treat-to-target dose titration scheme, injection s.c.
  Arms: B

SUMMARY:
This trial is conducted in the United States of America (USA) and Canada. The aim of this research is to compare the efficacy (reduction in HbA1c and blood glucose) and pulmonary safety (pulmonary function, chest x-rays) of mealtime inhaled insulin with subcutaneous insulin aspart both in combination with insulin determir in Type 1 Diabetes.

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* HbA1c less than or equal to 11%
* Body mass index (BMI) less than or equal to 40.0 kg/m2

Exclusion Criteria:

* Total daily insulin dosage more than 100 IU or U/day.
* Current smoking or smoking within the last 6 months
* Impaired hepatic or renal function
* Cardiac problems
* Uncontrolled hypertension
* Current proliferative retinopathy or maculopathy requiring acute treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2008-04-02 (Actual); Study Completion 2008-04-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 52 weeks

SECONDARY OUTCOMES:
Body weight | after 52 weeks
Antibodies | after 52 weeks
Hypoglycemia | For the duration of the trial
Insulin doses | For the duration of the trial
Pulmonary Function | For the duration of the trial
Fasting plasma glucose | after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (91):
- United States (81):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Tuscaloosa, Alabama
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, New Britain, Connecticut
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Merritt Island, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Lafayette, Indiana
  - Novo Nordisk Investigational Site, New Albany, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Scarborough, Maine
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Bloomington, Minnesota
  - Novo Nordisk Investigational Site, Duluth, Minnesota
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Tupelo, Mississippi
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Dover, New Hampshire
  - Novo Nordisk Investigational Site, Hampton, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (10):
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Gatineau
  - Novo Nordisk Investigational Site, Mississauga
  - Novo Nordisk Investigational Site, Penticton
  - Novo Nordisk Investigational Site, Red Deer
  - Novo Nordisk Investigational Site, St. John's
  - Novo Nordisk Investigational Site, Vancouver

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com